CLINICAL TRIAL: NCT01276873
Title: Clinical Variations and Pain Assessment in Newborns Submitted to Intratracheal Aspiration With Open and Closed System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Mavilde da Luz Gonçalves Pedreira, Associated professor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1094/09
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-12

CONDITIONS: Adverse Reaction to Systemic Agents
Keywords: Artificial Respiration; Suction; Pain; Nursing; Neonatology
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed System (Experimental): Application of Tracheal aspiration closed system, controlled by the use of Open system to tracheal aspiraiton.
  Interventions: Device: Tracheal aspiration close system

INTERVENTIONS:
Device: Tracheal aspiration close system — use of closed system in comparision to open system to tracheal aspiration of nweborns, analyzing pain and climical variations associated.
  Other Names: aspiration system; suctioning system; tracheal suctioning system

SUMMARY:
To compare clinical effects identified in infants undergoing intratracheal aspiration with open and closed systems and verify the presence and intensity of pain in newborns during intratracheal suction, according to the system applied.Clinical, randomized, controlled, and crossover study, performed at two neonatal intensive care units after approval by the ethics committee. The sample consisted of infants from zero to seven days of age, 26 weeks of gestational age, and the exclusion criteria were use of mechanical ventilation with high-frequency oscillatory, in use of inhaled nitric oxide, in the acute phase of circulatory failure, central nervous system disorders, without reactivity to stimulus, severe asphyxia, Apgar score less than three in the fifth minute, as well as, presence of chromosomal abnormalities and congenital malformations. After obtaining the informed consent from the responsible, children were randomly allocated into the experimental (CS) and control (OS) groups. The dependent variables of this study respiratory rate (RR), peripheral oxygen saturation (SatpO2), heart rate (HR), blood pressure (BP) and pain, as well as, of the complementary variables, were collected through observation, the Premature Infant Pain Profile (PIPP) scale application and medical records consultation. During the data collection the period of variables observation were: T1 (immediately before suctioning), T2 (during suctioning), T3 (immediately after) and T4 (10 minutes after). To the statistical analysis were applied Fisher exact test, McNemar, Binomial, Student t test, Wilcoxon and Mann Whitney, settling at 0.05 level of significance.

DETAILED DESCRIPTION:
Background: Patients who underwent tracheal intubation require intratracheal tube secretions sucking, and open system (OS) or closed system (CS) can be used, in order to preserve the tracheal tube permeability and an adequate ventilation and blood oxygenation. Respiratory and hemodynamic complications, as well as, presence of pain can be possibly experienced in newborns submitted to such procedure. Objectives: To compare clinical effects identified in infants undergoing intratracheal aspiration with OS or CS and verify the presence and intensity of pain in newborns during intratracheal suction, according to the system applied. Methods: Clinical, randomized, controlled, and crossover study, performed at two neonatal intensive care units after approval by the ethics committee. The sample consisted of infants from zero to seven days of age, 26 weeks of gestational age, and the exclusion criteria were use of mechanical ventilation with high-frequency oscillatory, in use of inhaled nitric oxide, in the acute phase of circulatory failure, central nervous system disorders, without reactivity to stimulus, severe asphyxia, Apgar score less than three in the fifth minute, as well as, presence of chromosomal abnormalities and congenital malformations. After obtaining the informed consent from the responsible, children were randomly allocated into the experimental (CS) and control (OS) gruops. The dependent variables of this study respiratory rate (RR), peripheral oxygen saturation (SatpO2), heart rate (HR), blood pressure (BP) and pain, as well as, of the complementary variables, were collected through observation, the Premature Infant Pain Profile (PIPP) scale application and medical records consultation. During the data collection the period of variables observation were: T1 (immediately before suctioning), T2 (during suctioning), T3 (immediately after) and T4 (10 minutes after). To the statistical analysis were applied Fisher exact test, McNemar, Binomial, Student t test, Wilcoxon and Mann Whitney, settling at 0.05 level of significance. Results: The studied groups did not show significant differences concerning the complementary variables. There were no statistically significant influences regarding the use of OS and CS of intratracheal suction in any of the dependent variables studied. Clinical consequences were observed with the use of both systems. It was demonstrated that immediately after intratracheal aspiration, the newborns had higher RR average in OS (58,4±9,6) group when compared to CS (56,2±5,9). Average values of SatpO2 were lower in OS (90,5±4,8) group compared to CS (91,6±4,6). Bradycardia was not verified in any group, however, there was a trend toward higher mean values of HR immediately after intratracheal aspiration, especially with OS (149,5±17,4) compared with the values identified before the procedure (143,2±18,1). There was low variation in the mean BP value in the two groups during the period of assessment, using both techniques. Regarding pain it was found that, with OS the average score was 7,9±4,4 and 6,5±3,8 with CS, demonstrating presence of mild to moderate pain. During the use of OS intratracheal aspiration higher pain scores (p=0,038) where verified in newborn females compared to males, this result was not observed when using CS. Conclusion: There was no statistically significant difference regarding the clinical implications, the presence and intensity of pain observed in ventilated newborns, according to the use of OS or CS to intratracheal aspiration.

ELIGIBILITY:
Inclusion Criteria:

* infants from zero to seven days of age.
* 26 weeks of gestational age.
* responsible concordance in participation

Exclusion Criteria:

* use of mechanical ventilation with high-frequency oscillatory.
* use of inhaled nitric oxide.
* acute phase of circulatory failure.
* central nervous system disorders.
* without reactivity to stimulus.
* severe asphyxia.
* Apgar score less than three in the fifth minute.
* Presence of chromosomal abnormalities and congenital malformations

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pain response to tracheal suction | 48 hours
  There were no statistically significant influences regarding the use of open (OS) or close system (CS) to intratracheal suction in this dependent variable. With OS the average score was 7,9±4,4 and 6,5±3,8 with CS, demonstrating presence of mild to moderate pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mavilde LG Pedreira, RN, PhD, Principal Investigator — Federal University of São Paulo; Jaqueline Cardoso, RN, Study Chair — Federal University of São Paulo; Ruth Guinsberg, MD, PhD, Study Chair — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Federtal university of São Paulo, São Paulo, São Paulo
  - Universidade Federal de São Paulo, São Paulo, São Paulo